CLINICAL TRIAL: NCT04996472
Title: A Developmental Framework For Linking Phonological and Morphosyntactic Sequential Pattern Rules in Developmental Language Disorder
Brief Title: A Framework For Linking Sequential Pattern Rules in DLD: Perception in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Father Flanagan's Boys' Home (Other)
Responsible Party: Principal Investigator, Lisa Goffman, Senior Scientist, Father Flanagan's Boys' Home
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2004574003R002 - Adults
Record Dates: First submitted 2021-07-22; First posted 2021-08-09 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Developmental Language Disorder; Speech Sound Disorder; Specific Language Impairment
MeSH Terms: conditions — Language Development Disorders; Speech Sound Disorder; Specific Language Disorder

STUDY DESIGN:
Intervention Model Description: Adults will complete case history, language history, and hearing screening. Participants will be randomly assigned to a condition, reflecting each of the 3 phonological patterns (Single Feature, OR, Family Resemblance). Randomization will occur within groups and will be generated a priori.
  Adults will participate in an experimental session, which includes exposure to the rule followed by a generalization test. A sub-group will participate in the Referential Study.
  Parents of the toddlers will fill out the expressive language MacArthur-Bates Communicative Development Inventory and also a case history. Toddlers will be assigned randomly to one of four conditions: OR condition with a referent; OR condition without a referent; Family Resemblance condition with a referent; Family Resemblance condition without a referent.
Who Masked: Participant
Masking Description: Participants will not be told which condition they are participating in. Investigators will know because of familiarity with the stimuli.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensitivity to phonological rules: Adults (Experimental): Arm 1: Single Feature Pattern; Arm 2: OR/Disjunction Pattern
  Interventions: Behavioral: Sensitivity to phonological rules: Adults
- Sensitivity to semantic category cues: Adults (Experimental): Arm 1. Referential cue during OR learning.
  Interventions: Behavioral: Sensitivity to semantic category cues: Adults

INTERVENTIONS:
Behavioral: Sensitivity to phonological rules: Adults — Assess whether adults are sensitive to different phonological patterns that are predicted to align with development of morphosyntax or the lexicon.
  Arms: Sensitivity to phonological rules: Adults
Behavioral: Sensitivity to semantic category cues: Adults — Assess whether adults show improved learning of OR or family resemblance rules when a semantic category cue is used.
  Arms: Sensitivity to semantic category cues: Adults

SUMMARY:
This broad aim of this clinical study is to assess the hypothesis that morphological and phonological deficits are linked by a broader deficit in sequential pattern learning. This hypothesis applies to learning in general, but is especially critical as an avenue for developing earlier assessments and more powerful interventions for children with developmental language disorder (DLD; AKA specific language impairment). Other populations, such as at-risk toddlers, may also benefit from this new approach.

DETAILED DESCRIPTION:
The developmental approach taken here combines what researchers already know about morpho-syntactic deficits in DLD with recent developments in the fields of linguistics and language acquisition. First, it is possible to divide phonological and morphological patterns into three pattern types (Single Feature, OR/Disjunction, Family Resemblance/Prototype), with these types having a long history of study in visual pattern learning. Importantly, children with DLD appear to have maximum difficulty with morpho-syntactic patterns of the OR type (e.g., regular past tense; add a "t" if the final consonant is voiceless OR a "d" if the final consonant is voiced). In contrast, studies using artificial grammars show that infants who are typically developing are highly adept at learning Single Feature and OR pattern types; Family Resemblance patterns may be weaker. Family resemblance patterns relate to similarity, and may be more closely tied to the lexicon than to grammar (e.g., beagles and terriers are similar and they are both dogs; the words "goat" and "boat" are similar). Typical adults are adept at Single Feature and Family Resemblance patterns, but appear to be, at least superficially, more like children with DLD in their performance on the OR pattern.

With these intriguing findings as a starting point, the proposed research links phonological and morphological sequence learning in children with developmental language disorder (DLD). In the studies focused on children, we ask if 4- to 6-year-olds who are typically developing as well as those with DLD (both with and without co-occurring speech sound deficits) and speech sound disorder (SSD; without co-occurring morpho-syntactic deficits) are sensitive to input examples that fit one of these three patterns. Our hypothesis is that, consistent with their long-documented morpho-syntactic deficit, children with DLD will have particular difficulty with the OR pattern. Consistent with their intact morpho-syntactic skills, children with SSD should show no deficits in the OR pattern, revealing a link between OR pattern learning, phonology, and morpho-syntax. Our endpoint measure is that children with DLD (both with and without an accompanying SSD) do not show sensitivity to the OR pattern, as measured by sound pattern (e.g., phonetic accuracy, syllable sequence stability) and motor learning (e.g., articulatory and acoustic variability) measures.

This hypothesis is assessed by indexing the learning trajectory across the training period and during generalization to new nonwords that are consistent or inconsistent with the training pattern. In the generalization phase, children are asked to name new novel words that are either consistent (i.e., that fit the training rule) or inconsistent (i.e., that do not fit the training rule) nonwords. It is predicted that children with TD and SSD, who are still in a period of language learning plasticity (they can still learn the sound patterns and grammar of a second language) will be sensitive to all three patterns. However, children with DLD (both with and without accompanying SSD) are predicted to show sensitivity to the family resemblance and single feature patterns, but not to the critical OR pattern-the one associated with sound pattern and grammatical learning, This would reveal an important connection between sound pattern and grammatical learning, which could lead to earlier diagnosis (phonological patterns emerge earlier than grammar) and to more general intervention practices that focus on sequential pattern learning rather than specific language goals may be efficacious.

A second aim explores whether the inclusion of a semantic subcategory cue facilitates learning the OR pattern. The hypothesis is that children with DLD (as well as typical adults) who initially are predicted to have the most difficulty with the OR pattern, will show increases in sensitivity following the addition of a semantic category cue (e.g., animals for the voiced consonant rule OR tools for the voiceless consonant rule). This result would be especially important for learners with DLD, as it may provide a pathway for intervention of a core learning deficit.

Critically, these studies are developmental in nature. In the adult component of this research, the investigators ask if adults are sensitive to input examples that fit one of these three patterns. Our hypothesis, based on previous findings from the Gerken lab, is that adults, like children with DLD, do not show sensitivity to the OR pattern. However, adults are sensitive to single feature and Family Resemblance patterns. Adults still learn words readily and are sensitive to family resemblance prototype relationships. For adults, perceptual measures index sensitivity. Similar to the children with typical development, DLD and SSD, the investigators explore whether the inclusion of a semantic subcategory cue facilitates learning the OR pattern in adults. The hypothesis is that all learners, including adults, will show increases in sensitivity following the addition of a semantic category cue (e.g., animals for voiced rule OR tools for voiceless rule). The findings from adults contribute to a dynamic developmental framework. Because of the dramatic developmental changes in sensitivity to phonological sound patterns and the presumed linkage of such patterns to morpho-syntax, the data from adults are essential in identifying the underlying mechanism(s) of DLD and to suggesting possible intervention strategies, such as employing semantic cues to the OR pattern and strengthening lexical organization.

From previous work, the investigators know that infants are sensitive to the OR rule. In the studies focused on toddlers, the investigators ask if dependence on the associatively organized lexicon can account for the infant-to-adult developmental changes observed for the OR pattern (which is not associatively organized) and thereby explores the possibility that children with DLD rely on their lexicons to compensate for their sequential pattern learning deficit. The hypothesis is that 20-month-old children, who are just entering a period of rapid vocabulary learning, will show increased sensitivity (based on looking time to words that are consistent vs. inconsistent within the training set) in the family resemblance condition when a visual referent (i.e., semantic cue) is added, but decreased sensitivity in the OR condition when a visual referent is added. These results will also be related to vocabulary size as reported on the CDI, with the prediction that robust patterns are smaller for children who received referents or who have smaller vocabularies for the OR pattern and greater for children who received referents or who have larger vocabularies for the family resemblance pattern. The results from toddlers, who are just entering a period of rapid vocabulary learning, provide an essential framework for understanding how different types of phonological patterns apply to lexical and morpho-syntactic learning, The results of the proposed study provide a critical developmental framework for identifying the underlying mechanism(s) of DLD. These findings will also lead to the development of intervention strategies, such as strengthening lexical organization, to support problematic aspects of sequential pattern learning.

ELIGIBILITY:
Inclusion Criteria:

Adults will have

* normal hearing
* will report no medical, educational, or developmental concerns in their case histories
* no history of speech, language, or hearing difficulties will be reported
* dominant exposure to English from infancy

Exclusion Criteria:

Participants will be excluded who have

* hearing impairment
* intellectual impairment
* autism
* significant motor impairment
* reported histories of developmental, speech, language, or hearing disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 933 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Adults' ability to learn different types of sound patterns measured by percent correct pattern identification at test | The assessment will be conducted immediately following the intervention
  After familiarization, adults will hear 16 test words (8 consistent and 8 inconsistent) and will judge whether each word was consistent or inconsistent with the alien language to which they were exposed. Learning is indexed based on judgment of consistent vs. inconsistent nonwords, with percent correct (saying "consistent" to truly consistent and "inconsistent" to truly inconsistent) as the dependent measure.
Adults' ability to learn different types of sound patterns with semantic cue measured by percent correct pattern identification at test | The assessment will be conducted immediately following the intervention
  After familiarization, adults will hear 16 test words (8 consistent and 8 inconsistent) and will judge whether each word was consistent or inconsistent with the alien language to which they were exposed. Learning is indexed based on judgment of consistent vs. inconsistent nonwords, with percent correct (saying "consistent" to truly consistent and "inconsistent" to truly inconsistent) as the dependent measure.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Goffman, PhD, Principal Investigator — Father Flanagan's Boys' Home
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - Boys Town Hospital, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided
It is the goal to share deidentified data on open science framework. Following the death of LouAnn Gerken, we are transferring the IRB.